CLINICAL TRIAL: NCT02573480
Title: Optimization Study of the Wraparound Care for Youth Injured by Violence Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of Funding
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Carolyn Snider, Associate Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2015:311
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Violence; Violence, Non-accidental; Physical Violence
Keywords: youth violence, intervention, emergency medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Wraparound Care (Experimental): Wraparound care initiated in the ED at the time of injury and continuing for approximately 1 year in the community.
  Interventions: Behavioral: Wraparound care

INTERVENTIONS:
Behavioral: Wraparound care — Wraparound care starts by linking an individual with a support worker who works with them to address risk factors and empower the individual to make positive choices. It not only includes connecting the youth with existing community resources such as education, employment, cultural services and substance counselling, it also helps build problem-solving skills, coping skills, and self-efficacy of the youth and family members. The support worker provides mentorship to the youth. Mentorship both teaches and emulates appropriate behaviours with respect to attitudes and behaviours associated with violence.

SUMMARY:
This study is an optimization study to evaluate how a wraparound program for youth who have been injured by violence helps to change violence related attitudes and beliefs, change individual risk factors for violence and reduce the risk of future injury due to violence. Wraparound care involves linking the youth with a support worker who will work with the youth to develop positive support networks and help them link with services that address risk factors towards future violence.

DETAILED DESCRIPTION:
In Canada, violence is the most common reason for youth (aged 12- 24) to visit an emergency department (ED) and the leading cause of hospitalization among males aged 20 to 24. Injury is a chronic, recurring disease. In Winnipeg, Canada, 20% of youth injured by violence visited the same ED in the next year with a repeat injury due to violence. Currently the standard of care for this vulnerable population is to discharge them from our EDs with no effort to prevent the next injury.

There are 5 components key to implementing wraparound care for youth who are at risk of violence. The 1st component is the establishment of a relationship between support worker and youth at the time of injury - i.e. during a teachable moment. The 2nd component is that the support worker has extensive "lived experience". Many youth affected by violence have been marginalized by society and have significant trust issues with figures of traditional power (i.e. doctors, social workers etc.). It is imperative that the support worker establish trust quickly and act as a role model. The 3rd component is that the care program is individualized for and by each youth. The support worker helps the youth to define their own goals and the steps required to achieve them. The 4th component is to provide trauma-informed care. Trauma-informed care is an approach used by caregivers that acknowledges the current and past traumas a person may have experienced and helps the person heal and build a sense of control over their lives. The final component is the opportunity to access community supports within their own culture.

ELIGIBILITY:
Inclusion Criteria:

1) Age 14 - 24, and 2) Presentation with an injury due to violence (defined as an injury inflicted by someone else and one caused by a gunshot wound, stab wound, blunt object, or bodily force).

Exclusion Criteria:

1) Unable to consent due to language or brain injury, 2) Sexual assault, 3) Child Abuse, 4) Self-Inflicted Injury, or 5) Transfer from hospital > 1 hr from Winnipeg, Canada

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Violence risk scores | 1 year post injury
  The Violence Risk Scale: Youth Version (YRS-YV) will be completed at intake and then again at 3 months, 6 months and 1 year. The total change score for each time period will be determined.

SECONDARY OUTCOMES:
Report risk/protective factors of youth injured by violence | Within 1 month post injury
  Many risk and protective factors such as education, employment, family, child protective services, access to health care, addictions, mental health, housing and interaction with the justice system have all been shown to be risk and in some cases protective (active education or employment) factors for violent injury among youth.
Prevalence of post-traumatic stress disorder (PTSD) among participants | Within 1 month post injury
  As indicated by PTSD Checklist - Civilian Version (PCL-C) and Structured Interview of Disorders of Extreme Stress (SIDES)
Prevalence of depression/mental health conditions among participants | Within 1 month post injury
  As indicated by the Patient Health Questionnaire (PHQ-9) Quick Depression Assessment and In addition to the PHQ-9, we will ask youth questions about previous mental health diagnoses to capture non-depression and PTSD diagnoses.
Prevalence of adverse childhood events (ACE) among participants | Within 1 month post injury
  As determined by scores on the Adverse Childhood Event questionnaire.
Prevalence of alcohol use disorder among participants | Within 1 month post injury
  As determined by scores on the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C).
Prevalence of (non-alcohol) substance use among participants | Within 1 month post injury
  As determined by scores on the Drug Use Questionnaire (DAST-10, Adolescent Version).
Intensity-of-care measurements | 1 year post-injury
  Based on a 3-part measurement developed by the Children's Hospital of Philadelphia (CHOP) as well as the more standard intensity measurements of total time used by San Francisco WrapAround care program and Healing Hurt People Program in Philadelphia. This measurement include: CHOP-method: 1) # of weeks receiving care, 2) # of needs addressed and 3) # of staff-client encounters; Standard Method: Total in-person contact time.
Rate of past year and post year visits to hospital for injury/substance use/mental health | 1 year pre and post injury
  Using ADT (Admissions, Diagnosis, Triage) and E-Triage and chart review, any visit to any ED in Winnipeg for intentional injury 1-year pre-index visit and 1-year post-index visit will be identified. Deaths due to violence will be identified using Vital Stats. Following the identification of a visit to the ED in the year pre and post the index injury (i.e. the injury at which time the youth participant was enrolled), a chart review at that hospital of that year will be completed.
Effect of EDVIP on resilience and post traumatic growth | 6 months and 1 year post injury
  Using Connor Davidson Resilience Scale and PostTraumatic Growth Injury, youth will be assessed for changes in resilience from baseline and posttraumatic growth at two time points.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Snider, MD, Principal Investigator — University of Manitoba
Locations (1):
- Winnipeg Health Sciences Centre, Winnipeg, Manitoba, Canada